CLINICAL TRIAL: NCT06339177
Title: Hemophagocytic Lymphohistiocytosis (HLH) Evaluation and Research of Clinical, ImmUnoLogic and TranscriptomE Study
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001899; 001899-I
Record Dates: First submitted 2024-03-29; First posted 2024-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-22

CONDITIONS: Lymphohistiocytosis, Hemophagocytic; Secondary Hemophagocytic Lymphohistiocytosis; Macrophage Activation Syndrome; Hyperinflammatory Syndromes
Keywords: Hemophagocytic Lymphohistiocytosis; HLH; Macrophage Activation Syndrome; MAS; Cytokine Storm Syndrome; Hyperinflammatory Syndrome; Hyperinflammation; Still's Disease; Hyperferritinemia; Immune Dysregulation
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Macrophage Activation Syndrome; Cytokine Release Syndrome; Arthritis, Juvenile; Hyperferritinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sHLH: Hemophagocytic lymphohistiocytosis (HLH) represents a clinical condition of persistent, dysregulated immune activation with unrelenting fevers, hyperferritinemia, and cytopenias, which lead to multiorgan failure and death.

SUMMARY:
Background:

Hemophagocytic lymphohistiocytosis (HLH) is a disease caused by disrupted immune function. People with HLH are prone to fevers and illnesses, which can be fatal. Some people develop a genetic form of this disease (pHLH), but researchers do not understand why some other people develop a nongenetic form (sHLH). They also do not have good ways to diagnose and treat sHLH.

Objective:

To learn about sHLH and why some people get it and others do not.

Eligibility:

Adults aged 18 years and older with sHLH.

Design:

Participants will be admitted to the study based on a review of their medical records. Those who join will have at least 3 clinical evaluations over 9 to 12 months. These may occur during an inpatient hospitalization if they require medical care or in the outpatient clinic.

Participants will also have a physical exam at each visit. Up to half a cup of blood will be drawn at each visit. Participants may also have their blood drawn by their own doctors, who will send the samples to the researchers. Researchers may also contact these participants by telephone or video calls.

The blood will be used for clinical tests as well as research. No new treatments will be administered as part of this study; however, standard medications and treatments may be recommended.

Participants may opt to continue their visits once a year for 3 more years. Participants may also opt for an extra clinial evaluation 1 week after starting a new treatment.

...

DETAILED DESCRIPTION:
Study Description:

The purpose of this multisite natural history study is to study the immunopathogenesis of secondary hemophagocytic lymphohistiocytosis (sHLH). This will include detailed longitudinal clinical and immunologic characterization of sHLH, as well as mechanistic studies evaluating inflammasome activation, cytotoxicity, and JAK-STAT signaling. Participants with sHLH will undergo clinical assessment and management along with three research blood draws with the option for additional blood draws at time points such as post-immunosuppressive treatment or treatment escalation and during longer-term follow-up. Participation may be in person or remote, with blood collected and processed locally then shipped to the NIH. Longitudinal clinical information will be recorded, and standard of care will be offered as needed.

Primary Objective:

To study the immunopathogenesis of sHLH from various etiologies including biomarkers, cellular phenotypes, and gene expression to determine mechanistic pathways that may be amenable to host-directed therapies.

Secondary Objectives:

* To prospectively and longitudinally characterize the predisposing conditions, clinical features, acute triggers, clinical labs, and outcomes of a cohort of individuals meeting sHLH criteria.
* To compare biomarkers and immune profiles between the classically defined sHLH subgroups (malignancy, autoimmune, immune-therapy, infectious-triggered, unknown etiology).
* To evaluate for novel immunologic subsets of sHLH with unsupervised analyses using a multi-omic approach, including single-cell transcriptomics and proteomics.
* To evaluate for rare, protein-altering variants in genes associated with cytotoxicity, inflammasome activation, or immunoregulation via (optional) co-enrollment in NIAID Centralized Sequencing protocol.

Primary Endpoint:

Identify immunologic mechanisms involved in the pathogenesis of sHLH from a variety of predisposing conditions.

Secondary Endpoints:

* Characterize the longitudinal clinical course of sHLH, including relapse rates and predictors of key clinical outcomes at one year after diagnosis.
* Identify differences in clinical and/or immunologic profiles between sHLH subgroups (malignancy, autoimmune, immune-therapy, infectious-triggered, unknown etiology).
* To evaluate for novel immunologic profiles in sHLH using multi-omic unsupervised analyses.
* Identify new genetic determinants of susceptibility to sHLH in the setting of different predisposing conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Aged 18 years or older.
* Established diagnosis of sHLH defined by meeting any published criteria, per Table 1:

  * Meeting the HLH-2004 criteria.
  * HScore of >168. For those without a bone marrow biopsy to evaluate for hemophagocytosis (worth 35 points in the criteria), HScore>134 will be used.
  * For those with underlying rheumatologic disease: meeting the 2016 American College of Rheumatology criteria for macrophage activation syndrome.
* Agree to storage and sharing of study data and biospecimens for future research use.

Table 1: Published Criteria for HLH

HLH-2004 Criteria:

Molecular diagnosis of HLH OR At least 5 of 8 below criteria:

* Fever (>38.4 Degrees Celcius)
* Splenomegaly
* Cytopenias affecting >=2 of 3 lineages: Hgb <9 g/dL, platelets <10^5/microliter, neutrophils <10^6/microliter
* Hypertriglyceridemia (>256 mg/dL) and/or fibrinogen <1.5 g/L
* Hemophagocytosis on biopsy
* Serum ferritin >=500 ng/mL
* Increased serum sCD25 (>2400 U/mL)
* Low or absent NK cell activity

HScore:

Known immunosuppression:

0 (no) or 18 (yes)

Temperature (degrees, Celsius):

0 (<38.4), 33 (38.4-39.4), 49 (>39.4)

Organomegaly:

0 (no), 23 (liver/spleen), 38 (both)

Number of cytopenias:

0 (1 lines), 24 (2 lines), 34 (3 lines)

Ferritin (ng/mL):

0 (<2000), 35 (2000-6000), 50 (>6000)

Triglycerides (mg/dL):

0 (<1.5), 44 (1.5-4), 66 (>4)

Fibrinogen (g/L):

0 (>2.5), 30 (<2.5)

AST (IU/mL):

0 (<30), 19 (>30)

Hemophagocytosis:

0 (no) or 35 (yes)

Cutoff value=169

ACR 2016-MAS Criteria:

A febrile patient with known or suspected sJIA is classified as having macrophage activation syndrome if the following criteria are met:

Ferritin >684 ng/mL

AND any 2 of the following:

* Platelets <=181,000/microliter
* AST >48 IU/mL
* Triglycerides >156 mg/dL
* Fibrinogen <=3.6 g/L

Abbreviations: ACR, American College of Rheumatology; AST, aspartate transaminase; Hgb, hemoglobin; HLH, hemophagocytic lymphohistiocytosis; MAS, macrophage activation syndrome; NK, natural killer, sJIA, systemic juvenile idiopathic arthritis.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Currently pregnant.
* Any condition that, in the judgment of the investigator, may put the participant at undue risk or make them unsuitable for participation in the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with active secondary HLH by meeting any published criteria. Hemophagocytic lymphohistiocytosis (HLH) represents a clinical condition of persistent, dysregulated immune activation with unrelenting fevers, hyperferritinemia, and cytopenias, which lead to multiorgan failure and death.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Identify immunologic mechanisms involved in the pathogenesis of sHLH from a variety of predisposing conditions. | Through end of study.
  To study the immunopathogenesis of sHLH from various etiologies including biomarkers, cellular phenotypes, and gene expression to determine mechanistic pathways that may be amenable to host-directed therapies.

SECONDARY OUTCOMES:
Prospectively define acute and longitudinal clinical profiles that predict key clinical outcomes. | Through end of study.
  To prospectively and longitudinally characterize the predisposing conditions, clinical features, acute triggers, clinical labs, and outcomes of a cohort of individuals meeting sHLH criteria.
Compare clinical and immune profiles between the classically defined HLH subgroups. | Through end of study.
  To compare biomarkers and immune profiles between the classically defined sHLH subgroups (malignancy, autoimmune, immune-therapy, infectious-triggered, unknown etiology).
Improve the understanding of the pathogenesis of sHLH. | Through end of study.
  To evaluate for novel immunologic subsets of sHLH with unsupervised analyses using a multi-omic approach, including single-cell transcriptomics and proteomics.
Characterize risk factors to identify populations at risk for developing sHLH. | Through end of study.
  To evaluate for rare, protein-altering variants in genes associated with cytotoxicity, inflammasome activation, or immunoregulation via (optional) co-enrollment in NIAID Centralized Sequencing protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Rocco, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and anonymized individual participant data collected in this study that underlie results in a publication will be made available after the end of the study by request.
Supporting Information: CSR
Time Frame: Upon completion of the protocol/upon publication.
Access Criteria: Data will only be available upon request, the PI will review and approve requests for data.

REFERENCES:
- [Background] Rocco JM, Laidlaw E, Galindo F, Anderson M, Sortino O, Kuriakose S, Lisco A, Manion M, Sereti I. Mycobacterial Immune Reconstitution Inflammatory Syndrome in HIV is Associated With Protein-Altering Variants in Hemophagocytic Lymphohistiocytosis-Related Genes. J Infect Dis. 2023 Jul 14;228(2):111-115. doi: 10.1093/infdis/jiad059. PMID 37040388
- [Background] Rocco JM, Laidlaw E, Galindo F, Anderson M, Rupert A, Higgins J, Sortino O, Ortega-Villa AM, Sheikh V, Roby G, Kuriakose S, Lisco A, Manion M, Sereti I. Severe Mycobacterial Immune Reconstitution Inflammatory Syndrome (IRIS) in Advanced Human Immunodeficiency Virus (HIV) Has Features of Hemophagocytic Lymphohistiocytosis and Requires Prolonged Immune Suppression. Clin Infect Dis. 2023 Feb 8;76(3):e561-e570. doi: 10.1093/cid/ciac717. PMID 36048425
- [Background] Shakoory B, Geerlinks A, Wilejto M, Kernan K, Hines M, Romano M, Piskin D, Ravelli A, Sinha R, Aletaha D, Allen C, Bassiri H, Behrens EM, Carcillo J, Carl L, Chatham W, Cohen JI, Cron RQ, Drewniak E, Grom AA, Henderson LA, Horne A, Jordan MB, Nichols KE, Schulert G, Vastert S, Demirkaya E, Goldbach-Mansky R, de Benedetti F, Marsh RA, Canna SW; HLH/MAS task force. The 2022 EULAR/ACR points to consider at the early stages of diagnosis and management of suspected haemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS). Ann Rheum Dis. 2023 Oct;82(10):1271-1285. doi: 10.1136/ard-2023-224123. Epub 2023 Jul 24. PMID 37487610
- [Background] Jordan MB, Allen CE, Greenberg J, Henry M, Hermiston ML, Kumar A, Hines M, Eckstein O, Ladisch S, Nichols KE, Rodriguez-Galindo C, Wistinghausen B, McClain KL. Challenges in the diagnosis of hemophagocytic lymphohistiocytosis: Recommendations from the North American Consortium for Histiocytosis (NACHO). Pediatr Blood Cancer. 2019 Nov;66(11):e27929. doi: 10.1002/pbc.27929. Epub 2019 Jul 24. PMID 31339233
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001899-I.html